CLINICAL TRIAL: NCT04308733
Title: Transcranial Direct Current Stimulation (tDCS) for Patients With Oro-pharyngeal Dysphagia Associated to Brainstem Stroke
Brief Title: tDCS for Dysphagia Associated to Brainstem Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Presidio Ospedaliero Garibaldi-Centro (Other)
Responsible Party: Principal Investigator, Domenico Antonio Restivo, Consutant Neurologist, Presidio Ospedaliero Garibaldi-Centro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Restivo Domenico
Record Dates: First submitted 2020-03-08; First posted 2020-03-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Active Comparator): 30 patients will be treated with real anodal tDCS over the contralateral pharyngeal motor cortex
  Interventions: Device: Anodal tDCS
- sham tDCS (Sham Comparator): 30 patients will be treated with sham tDCS over the contralateral pharyngeal motor cortex
  Interventions: Device: Anodal tDCS

INTERVENTIONS:
Device: Anodal tDCS — patients will be stimulated over the contralateral pharyngeal motor cortex with anodal tDCS (2mA, 20 minutes) for 4 consecutive days

SUMMARY:
The aim of the study is to investigate the effect of anodal transcranial direct current stimulation applied over the pharyngeal motor area in 60 dysphagic patients with acute isolated brainstem stroke. Thirty patients will undergo stimulation on the pharyngeal area contralateral to the side of brainstem lesion, and 30 patients will receive sham stimulation over the contralateral area, for 4 consecutive days. Patients will be re-evaluated after 4 consecutive days of stimulation. Primary outcome: The Penetration/Aspiration Scale after 4 consecutive days of stimulation. Secondary outcomes: changes in electromyographic parameters and pharyngeal cortical motor evoked potentials, changes in the Dysphagia Severity Rating Scale (DSRS), in the Functional Oral Intake Scale (FOIS), and in the "Dysphagia Limit Test", after 4 consecutive days of stimulation.

DETAILED DESCRIPTION:
Sixty consecutive patients with dysphagia associated to isolated acute (within the previous 24 hours) brainstem ischemic stroke satisfying the inclusion/exclusion criteria will be enrolled.

Swallowing evaluation Clinical evaluation comprises fiberoptic endoscopy that will be used for scoring the Penetration/Aspiration Scale. The Penetration/Aspiration Scale will be scored by two otolaryngologists and one neurologist blinded to the patient's study group allocation. Moreover, feeding status will be evaluated by the clinical "Dysphagia Severity Rating Scale", ranging from 0 (normal fluids, normal diet, and eating independently) to 12 (no oral fluids, no oral feeding). Moreover the "Functional Oral Intake Scale", ranging from 1 (nothing by mouth) to 7 (total oral diet with no restriction), and the "Dysphagia Limit Test", evaluating the amount of water that can be swallowed without piece-meal deglutition or clinical signs of aspiration, will be used in patient evaluation. Piecemeal deglutition will be evaluated both clinically and by means of electromyographic recordings from the mouth floor muscles. Moreover, simultaneous electromyographic/mechanographic recordings from the above mentioned muscles, as well as from cricopharyngeal muscle and from the thyroid cartilage will be also performed. The changes in cortico-pharyngeal excitability will be evaluated by recording motor evoked potentials from the pharyngeal muscles after transcranial magnetic stimulation.

Randomization: patients will be randomly assigned to either the active treatment (real) or sham groups according to a computer-generated list. Randomization will be stratified in order to match age, and severity of dysphagia.

Transcranial direct current stimulation: anodal transcranial direct current stimulation will be delivered through two 25-cm2 rectangular surface electrodes, with the active one placed over the "pharyngeal" area of the motor cortex contralateral to the side of brainstem lesion and the reference one on the contralateral supraorbital ridge. Furthermore, the electrodes will be fixed in their position using a set of adjustable rubber straps placed around the head. For the active intervention (the "real" stimulation group), current intensity will be slowly increased up to 2mA. This intensity will be maintained for 20 min before the stimulation will be slowly turned off over a 10-sec period. For the "sham" intervention, the current will be left on only for 30 sec, while the electrodes will be left in place for a further 20-min period. All patients will be evaluated at baseline, and after 4 consecutive days of stimulation.

ELIGIBILITY:
Inclusion Criteria:

* accepting to participating to the study
* age not < 18 years
* bulbar stroke occurring within the previous 24 hours

Exclusion Criteria:

* age < 18 years
* inability to give informed consent because of cognitive impairment
* stroke occurring over the previous 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Penetration Aspiration Scale (PAS) | Change from baseline PAS at 4 days
  PAS is an 8-point severity scale from 1 = no material enters the airways to 8 = material enters the airways, passes below the vocal folds in the absence of any effort to eject it.

SECONDARY OUTCOMES:
Functional Oral Intake Scale (FOIS) | Change from baseline FOIS at 4 days
  FOIS is a scale ranging from 1 (nothing by mouth) to 7 (total oral diet with no restriction)
Dysphagia Limit Test | Change from baseline "Dysphagia Limit Test" at 4 days
  The "Dysphagia Limit Test", evaluates the amount of water that can be swallowed without piece-meal deglutition or clinical signs of aspiration.
Pharyngeal (motor evoked potentials (MEPs) after Transcranial Magnetic Stimulation (TMS) | Change from baseline pharyngeal MEPs at 4 days
  the changes in amplitude of MEPs recorded from pharyngeal muscle after TMS over the pharyngeal contralateral motor cortex will be evaluated
electromyographic/cinematic evaluation of swallowing | Change from baseline electromyographic/cinematic parameters at 4 days
  Simultaneous electromyographic/cinematic recordings from mouth floor muscles, cricopharyngeal muscle and thyroid cartilage will be performed

CONTACTS AND LOCATIONS:
Locations (1):
- Domenico A. Restivo, Catania, Italy